CLINICAL TRIAL: NCT04538547
Title: Randomized Trial to Evaluate Accelerated Radiotherapy in the Management of Locally Advanced Carcinoma of Nasopharynx Using Rapid Arc Image Guided Radiotherapy
Brief Title: Randomized Trial to Evaluate Accelerated Radiotherapy in Locally Advanced Carcinoma of Nasopharynx
Acronym: EARN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Collaborators: Indian Council of Medical Research (Other Government)
Responsible Party: Principal Investigator, AMIT BAHL, ADDITIONAL PROFESSOR, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IEC-02/2019-1122
Record Dates: First submitted 2020-08-30; First posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-08

CONDITIONS: Carcinoma, Nasopharyngeal
Keywords: altered fractionation
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Accelerated Radiotherapy (Experimental): Accelerated Chemoradiotherapy followed by 3 cycles of Adjuvant chemotherapy. Patients will be treated with radiotherapy for 6 days per week from Monday to Saturday
  Interventions: Radiation: Accelerated Radiotherapy
- Non Accelerated Radiotherapy (Active Comparator): Concurrent Chemoradiotherapy followed by 3 cycles adjuvant chemotherapy. Patients will be treated with radiotherapy for 5 days per week from Monday to Friday.
  Interventions: Radiation: Non Accelerated Radiotherapy

INTERVENTIONS:
Radiation: Accelerated Radiotherapy — Accelerated Chemoradiotherapy followed by 3 cycles of Adjuvant chemotherapy. Patients will be treated with radiotherapy for 6 days per week from Monday to Saturday
  Arms: Accelerated Radiotherapy
Radiation: Non Accelerated Radiotherapy — Chemoradiotherapy followed by 3 cycles of Adjuvant chemotherapy. Patients will be treated with radiotherapy for 5 days per week from Monday to Friday
  Arms: Non Accelerated Radiotherapy

SUMMARY:
The present study is designed as a two arm randomized trial to evaluate the impact of accelerated radiotherapy delivered by image guided radiotherapy with rapid arc technique in carcinoma nasopharynx. The study will evaluate a pure acceleration schedule of 6 fractions per week with concurrent chemotherapy and without any radiotherapy dose escalation.The control arm will receive standard chemoradiotherapy using image guided radiotherapy with rapid arc technique.

DETAILED DESCRIPTION:
The study is designed as a two arm prospective randomized controlled trial which will be carried out in the Department of Radiotherapy and Otolaryngology at PGIMER, Chandigarh.

Inclusion criteria

1. Histopathologically proven non keratinizing nasopharangeal cancers.
2. Karnofsky performance status more than 70
3. Stage T3-4, N0-3 patients (as per AJCC 8th edition).
4. Patients willing for informed consent and regular follow up

Exclusion Criteria

1. Keratinizing squamous cell carcinoma
2. Age >70 years
3. Patients who have received previous chemoradiotherapy.
4. Patients with uncontrolled co- morbid conditions like hypertension , diabetes or any renal impairment

Randomization Patients will be randomized into the two study groups using computer generated randomization table given below.Total number of patients to be recruited will be 120 and will be divided into • Study Group A (N= 60): Accelerated Chemoradiotherapy followed by 3 cycles of Adjuvant chemotherapy. Patients will be treated with radiotherapy for 6 days per week from Monday to Saturday

• Control Group B (N=60) : Concurrent Chemoradiotherapy followed by 3 cycles adjuvant chemotherapy. Patients will be treated with radiotherapy for 5 days per week from Monday to Friday.

Treatment Protocol Clinical evaluation All patients enrolled in the study will undergo a full clinical examination including a complete head and neck check up Investigations All patients enrolled in the study will undergo the following investigations

1. Complete Haemogram, Liver Function test & Kidney Function Tests, Blood Sugar
2. Chest X Ray PA View
3. X Ray Soft tissue neck
4. ECG
5. CECT Head and Neck/ Contrast enhanced MRI head and neck
6. Biopsy from primary tumor and FNAC from neck nodes

RADIOTHERAPY Chemoradiotherapy treatment protocol For radiotherapy planning patients will be immobilized using S type thermoplastic cast & will undergo a planning CT scan with 3mm slice thickness. The images will be transferred to Eclipse treatment planning system. All patients will be planned with 6MV photons using 4 arcs with SIB Rapid Arc technique using the dose prescription given below.

PTV70: 70 Gy in 33 fractions PTV59.4 : 59.4 Gy in 33 fractions PTV50.4: 54 Gy in 33fractions Concurrent chemotherapy will be given using Cisplatin injection 40mg/m.sq weekly or 100mg/m.sq 3 weekly along with radiotherapy in both the groups. Patients will undergo will undergo a repeat treatment planning CT scan at the 16th radiotherapy fraction and will be evaluated for adaptive re-planning.

CHEMOTHERAPY Concurrent : Inj. CDDP 100mg/m2 D1 q 3weekly along with XRT

Adjuvant:

Inj. CDDP 80mg/ m2 D1 q 3 weekly x 3 cycles Inj. 5- FU 1gm/ m2 D1-4

Patients weight will be monitored weekly during treatment.patients will be reviewed at 16th fraction of treatment. Patients with a weight loss more than 10 % or a decrease of neck diameter by more than 10% will be evaluated for need for adaptive re-planning.Where indicated patients will be replanned .

Toxicity & Response Evaluation Patients will be evlautaed weekly for dermatological, mucositis,Dysphagia, haemtological ,gastrointestinal & constitutional toxicity using Common Terminology Criteria for adverse effects (CTCAE v3). Overall Response will be evaluated at end of treatment using Response evaluation criteria for solid Tumors (RECIST ).

Follow up All patients included in the study will be followed up 2 monthly intervals during the first year, at 3 monthly intervals during the 2-3 years and 6 monthly intervals thereafter. At each visit a full clinical examination, toxicity grading and disease status will be evaluated.

Statistics Assuming a significance level of 0.05 and power of 80% a minimum of 110 patients need to be recruited to detect a difference of about 25% in failure free survival including a drop out rate of 10%.For statistical analysis data will be entered into SPSSv 20.Treatment toxicity will be compared between the treatment groups using independent 't' test. Pearson correlation test and logistic regression analysis will be used to evaluate prognostic variables.Survival analysis will be done using Kaplan Meir analysis. A p value <0.05 will be considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically proven non keratinizing nasopharangeal cancers.
2. Karnofsky performance status more than 70
3. Stage T3-4, N0-3 patients (as per AJCC 8th edition).
4. Patients willing for informed consent and regular follow up

Exclusion Criteria:

1. Keratinizing squamous cell carcinoma
2. Age >70 years
3. Patients who have received previous chemoradiotherapy.
4. Patients with uncontrolled co- morbid conditions like hypertension , diabetes or any renal impairment

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-09-16 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
To compare acute treatment related toxicity between the two study groups | Within 90 days of completion of treatment
  Patients under study will be monitored for acute toxicity using CTCAEv3
To compare overall response rates between the two study group | At 1 year follow up
  Overall survival will be compared between the study and control group at end of study

CONTACTS AND LOCATIONS:
Overall Officials: AMIT BAHL, MD, Principal Investigator — PGIMER CHANDIGARH INDIA
Locations (1):
- Post Graduate Institute of Medical Education and Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee AW, Sze WM, Yau TK, Yeung RM, Chappell R, Fowler JF. Retrospective analysis on treating nasopharyngeal carcinoma with accelerated fractionation (6 fractions per week) in comparison with conventional fractionation (5 fractions per week): report on 3-year tumor control and normal tissue toxicity. Radiother Oncol. 2001 Feb;58(2):121-30. doi: 10.1016/s0167-8140(00)00312-1. PMID 11166862
- [Background] Blanchard P, Lee A, Marguet S, Leclercq J, Ng WT, Ma J, Chan AT, Huang PY, Benhamou E, Zhu G, Chua DT, Chen Y, Mai HQ, Kwong DL, Cheah SL, Moon J, Tung Y, Chi KH, Fountzilas G, Zhang L, Hui EP, Lu TX, Bourhis J, Pignon JP; MAC-NPC Collaborative Group. Chemotherapy and radiotherapy in nasopharyngeal carcinoma: an update of the MAC-NPC meta-analysis. Lancet Oncol. 2015 Jun;16(6):645-55. doi: 10.1016/S1470-2045(15)70126-9. Epub 2015 May 6. PMID 25957714
- [Background] Lacas B, Bourhis J, Overgaard J, Zhang Q, Gregoire V, Nankivell M, Zackrisson B, Szutkowski Z, Suwinski R, Poulsen M, O'Sullivan B, Corvo R, Laskar SG, Fallai C, Yamazaki H, Dobrowsky W, Cho KH, Beadle B, Langendijk JA, Viegas CMP, Hay J, Lotayef M, Parmar MKB, Auperin A, van Herpen C, Maingon P, Trotti AM, Grau C, Pignon JP, Blanchard P; MARCH Collaborative Group. Role of radiotherapy fractionation in head and neck cancers (MARCH): an updated meta-analysis. Lancet Oncol. 2017 Sep;18(9):1221-1237. doi: 10.1016/S1470-2045(17)30458-8. Epub 2017 Jul 27. PMID 28757375